CLINICAL TRIAL: NCT02790593
Title: A Randomised Controlled Clinical Trial Comparing the Effectiveness of Bandaging Compared to the Juxta-CuresTM Device in the Management of People With Venous Ulceration: Feasibility Study
Brief Title: Juxta-CuresTM Versus Bandaging for Venous Ulcers
Acronym: Juxta-Cures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colchester Hospital University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Juxta-CuresTM (2016/006)
Record Dates: First submitted 2016-05-03; First posted 2016-06-06 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Venous Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juxta-Cures™ (Experimental): Patients randomised to the Juxta-Cures™ device. These patients will also have pressure monitoring using the PicoPress device, and ulcer imaging and surface area measurement using the Silhouette system.
  Interventions: Device: Juxta-Cures™; Device: PicoPress®; Device: Silhoutte® 3D wound imaging system
- Standard compression (Active Comparator): Patients randomised to standard compression. These patients will also have pressure monitoring using the PicoPress device, and ulcer imaging and surface area measurement using the Silhouette system.
  Interventions: Device: Standard Compression; Device: PicoPress®; Device: Silhoutte® 3D wound imaging system

INTERVENTIONS:
Device: Juxta-Cures™ — Juxta-CURES™ is an adjustable compression device, which may be used as a secondary dressing for the treatment of open venous stasis ulcers. It is an inelastic wrap around device with a Built-In-Pressure System™, which allows patients to easily and accurately apply pressure to their own leg and adjust it throughout the day.
  Arms: Juxta-Cures™
Device: Standard Compression — Compression bandaging
  Arms: Standard compression
Device: PicoPress® — Pressure monitoring to be done at time of bandage application and removal for both arms of the study.
Device: Silhoutte® 3D wound imaging system — Photographic imaging system to measure wound surface area and depth. Picture to be taken at each appointment. This intervention is for both arms of the study.

SUMMARY:
Venous ulceration is a major burden on the NHS. Current treatment involves bandaging therapy which is replaced on a once or twice weekly basis. The Juxta-CuresTM device offers an alternative solution for the long-term treatment of patients with venous ulceration. This is a removable adjustable device with an inbuilt pressure monitor. The aim of this study is to determine whether the Juxta-Cures™ device provides at least equivalent ulcer healing for patients with venous ulceration compared to bandaging. Secondary outcome measures include whether the Juxta-Cures™ device improves patient compliance and quality of life compared to bandaging, and whether the Juxta-Cures™ device is cost effective compared to bandaging.

DETAILED DESCRIPTION:
Participants with lower leg ulceration will be identified at consultant or nurse-led clinics. They will be assessed by their clinician, and identified as having a likely venous ulcer. Participants undergoing current leg ulcer management of any type may be considered for this trial. At this stage participants will be given the most recent version of the patient information sheet, given appropriate initial treatment as determined by their clinician (simple dressings, or compression bandaging if appropriate), and booked for venous and arterial duplex as well as ABPI which will be undertaken within 10 +/- 4 days. The patient will then be reviewed in 10 days +/- 4 days at venous ulcer clinic to discuss any queries regarding the trial with their clinician. Informed consent will be obtained from all participants at this point if appropriate, and the patient will be randomised, (a minimum of 24 hours will be required for the patient to read the information prior to giving informed consent).

Following randomisation the participant will be reviewed in the leg ulcer clinic on a 10 +/- 4 days basis whereby pressure monitoring will be conducted using the PicoPress® (Microlan Italia, Padua, Italy), dressings will be changed and ulcer measured with standard 1cm squared grids, and the Silhoutte® 3D wound imaging system (ARANZ Medical Ltd, Christchurch, New Zealand). Participants will also submit their daily use and pressure diary. The type of dressings applied will also be recorded as well as length of appointment.

50 participants will be recruited (aim for study duration of 12-18 months) from a consultant or nurse-led clinic at Colchester Hospital and associated outlying clinics, and participants randomised to receive either compression bandages or Juxta-Cures™ (bilateral participants will be allocated a single treatment, rather than randomisation of individual limbs). Patients with 'wet' ulcers may receive absorbent dressings under Juxta-Cures™ or compression bandaging during the study period, which will be recorded on the weekly data collection for cost analysis purposes.

At baseline, 1 month, 3 months and 6 months all participants will complete health related quality of life questionnaires. The disease specific VEINESqol/sym, and generic Euroqol-5D-5L surveys will be used, and received positive feedback regarding their content at the patient focus group.

The planned study period for the randomised-control trial is 24 weeks for each participant, but 1 year in total for patient recruitment and analysis.

This study is a feasibility study therefore has not been powered. Following this study the investigators aim to undertake a multi-centre study in collaboration with the Vascular and Endovascular Research Network (VERN), powered to venous ulcer healing at 90% power, using the results of this feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Active venous ulcer for >2 weeks but <1 year

  * 1cm squared surface area
  * Venous incompetence confirmed by clinical assessment and duplex ultrasound scan
  * No evidence of arterial disease (Arterial Duplex or Ankle Brachial Pressure Index >0.9)
  * Patients able to complete trial procedures
  * Patients with a life expectancy of greater than 1 year

Exclusion Criteria:

* Age less than 18 years
* Significant arterial disease (Ankle Brachial Pressure Index <0•9 or evidence on Arterial Duplex)
* Acute Deep Vein Thrombosis
* Patient unable or unwilling to have high compression (30mmHg minimum)
* Patients with dexterity insufficiency of hands
* Patients with peripheral neuropathy
* Leg ulcers of another underlying cause
* Leg ulcers of greater than 1 year duration
* Patients unable or unwilling to provide written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients for this study per 100,000 population | 1 year
Percentage of eligible patients accepted for randomisation | 1 year
Patient compliance with trial protocol, measured as days without compression in trial period | 1 year
Percentage of patients completing study | 1 year (to run entire study including patient recruitment, with each patient enrolled for 6 months)
  Those patient completing 6 months of treatment or ulcer healing from all entering study.

SECONDARY OUTCOMES:
Change in ulcer diameter measured by cm squared. | 1 year
Change in ulcer diameter measured by cm cubed. | 1 year
Change in ulcer diameter measured by percentage. | 1 year
Ulcer healing rate | 1 year (to run entire study including patient recruitment, with each patient enrolled for 6 months)
  Percentage of patients with healed ulcers at 6 months
Patient quality of life measured by EuroQol-5D-5L | 1 year
  Aim to determine differences in quality of life using each device
Patient quality of life measured by VEINESqol/sym | 1 year
  Aim to determine differences in quality of life using each device
Cost effectiveness | 1 year
  Total cost of treatment in each arm of the study, measured in pounds sterling
Pressure consistency | 1 year
  Monitor of pressure at bandage application and removal to determine which arm of the trial delivers more consistent pressure

CONTACTS AND LOCATIONS:
Overall Officials: Adam Howard, Principal Investigator — Colchester Hospital NHS Foundation Trust; Philip Stather, Principal Investigator — Colchester Hospital NHS Foundation Trust
Locations (1):
- NHS Trust, Colchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No